CLINICAL TRIAL: NCT06738992
Title: Safety and Effectiveness of Early Aspirin Administration After Mitral Valve Repair: a Prospective, Non-inferiority, Randomized Controlled Clinical Trial Protocol
Brief Title: Safety and Effectiveness of Early Aspirin Administration After Mitral Valve Repair
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KY2024-767-02
Record Dates: First submitted 2024-12-06; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Mitral Valve Repair Surgery
Keywords: mitral valve repair surgery; Warfarin; Aspirin
MeSH Terms: interventions — Aspirin; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Warfarin Group (Active Comparator): Anticoagulation therapy was initiated on the second day after surgery, starting at 4.5 mg once nightly, with adjustments made based on changes in the INR value.
  Interventions: Drug: Warfarin
- Aspirin Group (Experimental): Antiplatelet therapy was initiated on the second day after surgery with oral administration of Aspirin Enteric-coated Tablets (Bayer Aspirin) at a dose of 100 mg once daily.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — Antiplatelet therapy was initiated on the second day after surgery with oral administration of Aspirin Enteric-coated Tablets (Bayer Aspirin) at a dose of 100 mg once daily.
  Arms: Aspirin Group
Drug: Warfarin — Anticoagulation therapy was initiated on the second day after surgery, starting at 4.5 mg once nightly, with adjustments made based on changes in the INR value.
  Arms: Warfarin Group

SUMMARY:
This study compares the efficacy and safety of two different antithrombotic drugs, warfarin and aspirin, in early application after mitral valve repair (MVRep). The objective is to verify whether the type of antithrombotic therapy affects clinical outcomes and the incidence of thromboembolic and bleeding complications within 3 months after MVRep, and to provide safe and effective antithrombotic treatment options for patients undergoing MVRep.

DETAILED DESCRIPTION:
Patients were randomly assigned in a 1:1 ratio to two groups: the Warfarin Group and the Aspirin Group.

Warfarin Group: Anticoagulation therapy was initiated on the second day after surgery, starting at 4.5 mg once nightly, with adjustments made based on changes in the INR value.

Aspirin Group: Antiplatelet therapy was initiated on the second day after surgery with oral administration of Aspirin Enteric-coated Tablets (Bayer Aspirin) at a dose of 100 mg once daily.

For all patients, antithrombotic therapy was continued for at least 3 months post-surgery. Patients were scheduled for outpatient visits at 1, 4, 8, and 12 weeks following the surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years and above, but not exceeding 85 years;
* Patients who have successfully undergone mitral valve plasty with implantation of a mitral annuloplasty ring, with the option to undergo concurrent tricuspid valve plasty, atrial septal defect repair, or myxoma resection;
* Patients with preoperative electrocardiogram (ECG) showing sinus rhythm;
* Alternatively, patients with preoperative ECG showing atrial fibrillation (AF) rhythm, but who are male with a CHA2DS2-VASc-60 score of 0 or female with a score of 1; for patients with a CHA2DS2-VASc-60 score exceeding the aforementioned values but who have successfully converted to sinus rhythm following concurrent radiofrequency catheter ablation for AF;
* Patients who voluntarily participate in this study, have signed a written informed consent form, and are willing to comply with follow-up procedures.

Exclusion Criteria:

* Patients with contraindications to any of the following medications: heparin, warfarin, or aspirin;
* Patients who have undergone artificial valve replacement at other valve positions;
* Patients with a high risk of bleeding (including active bleeding, platelet count <50×10^9/L, hemoglobin <8.0 g/dL, history of cerebral hemorrhage, active peptic ulcer, or history of gastrointestinal bleeding within the last 3 months);
* Patients with acute coronary syndrome within the last month;
* Patients with symptomatic stroke within the last 3 months;
* Patients with renal insufficiency and a creatinine clearance rate <30 mL/min; Dialysis patients;
* Patients with moderate or severe hepatic impairment or liver disease with coagulation dysfunction: Child-Pugh score greater than B or bilirubin greater than or equal to 2 times the upper limit of normal (ULN) as defined by the center, and alanine aminotransferase (ALT), aspartate aminotransferase (AST), or serum alkaline phosphatase (ALP) levels greater than or equal to 3 times the ULN as defined by the center;
* Patients with active malignant tumors;
* Patients who are planned to undergo surgical intervention or treatment (including endoscopy) during the trial period that requires discontinuation of anticoagulants;
* Pregnant or lactating women, or fertile individuals unwilling or unable to use effective contraceptives;
* Patients who have participated in any drug clinical trial within the last 6 months prior to screening;
* Patients who refuse to undergo follow-up;
* Patients deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical thromboembolic events | From enrollment to the end of treatment at 12 weeks
  Clinical thromboembolic events are defined as stroke, myocardial infarction, symptomatic valve thrombosis, systemic embolism, deep venous thrombosis, or pulmonary embolism.
Asymptomatic intracardiac thrombosis | From enrollment to the end of treatment at 12 weeks
  Asymptomatic intracardiac thrombosis is defined as subclinical leaflet thrombosis or intracavitary thrombus detected by cardiac computed tomography (CT) or echocardiography within 12 weeks postoperatively. Subclinical leaflet thrombosis is defined as leaflet thickening with reduced leaflet motion and at least moderate (reduction >50%) valve area obstruction, demonstrated by cardiac CT, with a lesser degree of leaflet thinning.
Death due to cardiovascular causes or thromboembolic events | From enrollment to the end of treatment at 12 weeks
Major bleeding | From enrollment to the end of treatment at 12 weeks
  Fatal bleeding; and/or symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular, or pericardial or intramuscular bleeding with compartment syndrome; and/or bleeding resulting in a decrease in hemoglobin level by 3.0 g/dL。

SECONDARY OUTCOMES:
postoperative length of hospital stay | From enrollment to the end of treatment at 12 weeks
  from the day of surgery to the first discharge
International normalized ratio at the time of thromboembolic or bleeding events | From enrollment to the end of treatment at 12 weeks
CHA2DS2-VASc scores | From enrollment to the end of treatment at 12 weeks
  The CHA2DS2-VASC score is a risk stratification tool for assessing the likelihood of stroke in patients with non-valvular atrial fibrillation. The maximum score is 9, and the minimum score is 0.A lower CHA2DS2-VASC score is generally considered better.
HAS-BLED scores | From enrollment to the end of treatment at 12 weeks
  The HAS-BLED score is a scoring system used to predict the risk of bleeding in patients with atrial fibrillation undergoing anticoagulant therapy. Its full name is the "Hemorrhagic risk in Atrial fibrillation patients on anti-coagulation therapy using European League Against Rheumatism (EULAR) criteria, Bleeding Academic Research Consortium (BARC) definitions" score system, often abbreviated as HAS-BLED.The maximum score is 9, and the minimum score is 0.A lower HAS-BLED score is generally considered better.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Baseline Characteristics, Outcome Measures, Adverse Events and so on
Supporting Information: CSR